CLINICAL TRIAL: NCT06367478
Title: Evaluation of Acquisition Parameters and Stimulation to Obtain Different Neurophysiological Responses
Brief Title: Evaluation of Nerve Conduction Study
Acronym: SPEMG
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: SPEMG
Record Dates: First submitted 2024-03-29; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Nerve Condition; Health, Subjective

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the investigators study different modality to obtain nerve evoked reponses. They use different parameters of acquisition and stimulation and they compare amplitude and latency of nerve conduction response

ELIGIBILITY:
Inclusion Criteria:

* absence of previous nervous pathologies

Exclusion Criteria:

* nerve disease
* diabetes
* polyneuropathy

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: healthy subjects
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2024-10-22 (Estimated)

PRIMARY OUTCOMES:
best amplitude of nerve conduction study | baseline and after 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico of Milan, Milan, Italy